CLINICAL TRIAL: NCT05720832
Title: Technology-Based Social-Support Intervention Program for Reducing Psychosocial Burden in Prostate Cancer Patients: A Proof-of-Feasibility Pilot Study
Brief Title: Feasibility of Technology-Based SSIP in Prostate Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wings Health AG (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-02095
Record Dates: First submitted 2023-01-16; First posted 2023-02-09 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer; Psychosocial Stressor
Keywords: prostate cancer; social support; mental health; psychosocial intervention; pilot study
MeSH Terms: conditions — Prostatic Neoplasms; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate Cancer Patients and their Supporters (Experimental): The WINGS smartphone application is being tested on prostate cancer patients for the first time in this pilot study. It provides easy access to prostate cancer-related information and simplifies networking with supporters, such as family and friends. The WINGS smartphone application can be easily downloaded to a personal smartphone via Google Play or the App Store and can be used at any time from home or on the go.
  In addition, the WINGS smartphone application also provides supporters, such as family members and friends of prostate cancer patients with easy access to prostate cancer-related information. Moreover, it helps them to support prostate cancer patients by facilitating joint activities, tailored to the needs of the patient.
  Interventions: Other: WINGS-IP1 Smartphone Application

INTERVENTIONS:
Other: WINGS-IP1 Smartphone Application — The technology-based SSIP ("WINGS") offers disease-related information and builds up social inner circles between patients, their friends, and family members while facilitating to organize, perform, and enjoy activities and content.
  Other Names: technology-based social-support intervention program

SUMMARY:
The goal of this pilot study is to assess the perceived usability of a smartphone application called WINGS targeting psychosocial distress and well-being in prostate cancer patients and their social network. The main questions it aims to answer are:

* How do prostate cancer patients and their social network rate the usability of the technology-based social-support intervention program smartphone application?
* Do symptoms of prostate cancer patients improve after using the WINGS smartphone application?
* Does the burden of prostate cancer patients social network decrease after using the WINGS smartphone application? Participants will be asked to use the WINGS smartphone application over the period of eight to twelve weeks and fill in questionnaires before, during, and after this time.

DETAILED DESCRIPTION:
There is still little knowledge about how smartphone apps can improve the quality of life in prostate cancer patients. Hence, the investigators are interested in finding out whether the simplified access to information and planning of activities increases the perceived social support in prostate cancer patients and ultimately improves their quality of life.

The duration of the study is approximately three months per participant. The WINGS smartphone application can be used from home and questionnaires can be completed online. Participants are therefore not required to be present at the University Hospital Basel during the entire course of the present study.

The investigators plan to recruit a total of 30 prostate cancer patients at the University Hospital Basel and 0-10 supporters (family members and friends) per prostate cancer patient. All study participants will have access to the regular treatment services of the University Hospital Basel.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written consent
* Male;
* ≥ 18 years of age;
* Sufficient knowledge of German language;
* Confirmed diagnosis of prostate carcinoma;
* Successfully completed prostatectomy with "Da Vinci®" method;
* Willingness to use the WINGS-IP1 Smartphone Application (technology-based SSIP);
* In possession of a smartphone on which the WINGS-IP1 Smartphone Application V1.0 can be installed (required operating systems: iOS 12.1 or newer, Android 7.0 or newer);
* Access to the Internet with smartphone;
* Ability to operate a smartphone;

Exclusion Criteria:

* Previous enrolment in the current investigation;
* Current diagnosis of severe mental disorder, namely bipolar disorder, schizophrenia, personality disorder;
* Simultaneous participation in any other clinical trial, hospital program, or psychosocial intervention targeting similar concepts (e.g., mental wellbeing, social support, sexuality, etc.);
* Receiving any current treatment for mental disorder (psychotherapy and/or medication) apart from already existing long-lasting therapies (≥ 6 months);

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Subjective Usability | post-intervention (after 8 weeks)
  Primary outcome is prostate cancer patients' perceived usability of the WINGS-IP1 Smartphone Application measured by the German version of the 'Intervention Usability Scale' (IUS, [Lyon et al., 2021]). This scale was adapted from the 'System Usability Scale' (SUS, [Brooke, 1996]), a widely used self-reported scale to assess usability of digital systems, mobile applications, devices, and websites (see Kaya et al., 2019; Klug, 2017; Usability.gov, 2013). The SUS is composed of 10 items, assessed on a five-point Likert-scale, ranging from 0 = "strongly disagree" to 4 = "strongly agree" (Brooke, 1996). This scale will be completed by prostate cancer patients and their supporters.

SECONDARY OUTCOMES:
Subjective Usability Follow-up | follow-up (after 12 weeks)
  Primary outcome is prostate cancer patients' perceived usability of the WINGS-IP1 Smartphone Application measured by the German version of the 'Intervention Usability Scale' (IUS, [Lyon et al., 2021]). This scale was adapted from the 'System Usability Scale' (SUS, [Brooke, 1996]), a widely used self-reported scale to assess usability of digital systems, mobile applications, devices, and websites (see Kaya et al., 2019; Klug, 2017; Usability.gov, 2013). The SUS is composed of 10 items, assessed on a five-point Likert-scale, ranging from 0 = "strongly disagree" to 4 = "strongly agree" (Brooke, 1996). This scale will be completed by prostate cancer patients and their supporters.
Change in Mental Burden Related to Medical Condition | pre-intervention (T1), post-intervention (8 weeks after T1), follow-up (12 weeks after T1)
  In order to assess change mental burden related to medical condition the investigators will use the German version of the 'Mental Health Component Summary Score' of the 'Short Form-36 Version 1'(SF-36, [Ware, 2000]). The SF-36 is a validated, self-report instrument consisting of 36 items rated on five-choice response scales. The possible score ranges from 0 to 100 points, whereby 0 points represent the greatest possible health restriction and 100 points represent no health restriction at all. This scale will only be completed by prostate cancer patients.
Change in Depressive Symptoms | pre-intervention (T1), post-intervention (8 weeks after T1), follow-up (12 weeks after T1)
  The investigators will use the German version of the 'Patient Health Questionnaire' with 8 items (PHQ-8) to assess the severity of depressive symptoms in prostate cancer patients (Kroenke et al., 2009; Kroenke & Spitzer, 2002). The last criteria had been excluded as it assesses suicidal or self-injurious thoughts, which investigators will not be able to address adequately within the context of the proposed study. Prostate cancer patients and their supporters will be asked to indicate how often they experienced a depressive symptom in the past two weeks (Kroenke et al., 2009). They rate these symptoms on a four-point Likert-scale ranging from 0 = "not at all," 1 = "several days," 2 = "more than half the days," to 3 = "nearly every day". The PHQ-8 demonstrated acceptable internal consistency with Cronbach's α = 0.82 (Pressler et al., 2011).
Change in Anxiety | pre-intervention (T1), post-intervention (8 weeks after T1), follow-up (12 weeks after T1)
  The investigators will implement the German version of the seven item 'General Anxiety Disorder Scale' (GAD-7) to assess the presence of generalized anxiety disorder, social phobia, panic disorder, and post-traumatic stress disorder (Spitzer et al., 2006; Staples et al., 2019). Prostate cancer patients and their supporters rate items on a four-point Likert-scale ranging from 0 = "not at all," 1 = "several days," 2 = "more than half the days," to 3 = "nearly every day", based on their symptoms in the last two weeks. The GAD-7 showed acceptable discriminative validity (AUCs between 0.74 and 0.75, ps < 0.001) and good test-retest reliability (r = 0.83) and internal consistency with Cronbach's α = 0.88 (Staples et al., 2019).
Daily Symptom Trajectories: Depressive Symptoms and Anxiety | daily assessment during 8 week intervention phase
  In order to measure daily fluctuations of depressive symptoms and anxiety during the eight-week intervention phase, the investigators will implement the 'Patient Health Questionnaire' (PHQ-4) which consists of the PHQ-2 (Kroenke et al., 2003) and the 'General Anxiety Disorder Scale' (GAD-2, [Staples et al., 2019]) as Ecological Momentary Assessment (EMA, [Stone et al., 1999]). Both measures will be adapted in accordance with procedures of Bauer and colleagues (2018) to adjust instructions and Likert-scales to daily assessments. This scale will only be completed by prostate cancer patients.
Change in Perceived Social Stigma | pre-intervention (T1), post-intervention (8 weeks after T1), follow-up (12 weeks after T1)
  In the proposed study the investigators will assess prostate cancer patients perceived stigma using the German version of the 'Social Impact Scale' (SIS-D) with 24 items (Fife & Wright, 2000). The SIS-D has been previously used to measure stigma in cancer patients and covers four dimensions, namely social rejection, internalised shame, social isolation, and financial insecurity. All items are answered on a 4-point Likert scale from 1 ("strongly disagree") to 4 ("strongly agree"). This scale will only be completed by prostate cancer patients.
Change in Perceived Social Support | pre-intervention (T1), post-intervention (8 weeks after T1), follow-up (12 weeks after T1)
  To assess prostate cancer patients' perceived social support, the investigators will use the German version of the 'Oslo Social Support Scale' (OSSS-3, [Dalgard et al., 2006; Kocalevent et al., 2018]). The OSSS-3 is a very brief, three-item scale. In addition to pre- and post-intervention assessment, the investigators will also measure the OSSS-3 weekly, to assess fluctuations in perceived social support. The sum score ranges from 3 to 14, with high values representing strong levels and low values representing poor levels of social support. This scale will only be completed by prostate cancer patients.
Weekly Change in Perceived Social Support | weekly assessment during 8 week intervention phase
  To assess prostate cancer patients' perceived social support, the investigators will use the German version of the 'Oslo Social Support Scale' (OSSS-3, [Dalgard et al., 2006; Kocalevent et al., 2018]). The OSSS-3 is a very brief, three-item scale. In addition to pre- and post-intervention assessment, the investigators will also measure the OSSS-3 weekly, to assess fluctuations in perceived social support. The sum score ranges from 3 to 14, with high values representing strong levels and low values representing poor levels of social support. This scale will only be completed by prostate cancer patients.
Change in Somatic Symptom Disorder | pre-intervention (T1), post-intervention (8 weeks after T1), follow-up (12 weeks after T1)
  The investigators will assess somatic symptom disorder using the 'Somatic Symptom Disorder-B Criteria Scale' (SSD-12) composed of 12 items (Toussaint et al., 2016). These subscales are divided into three psychological subscales including cognitive aspects, affective aspects, and behavioural aspects. All items are answered on a 5-point Likert scale from 1 ("never") to 4 ("very often"). This scale will only be completed by prostate cancer patients.
Change in Symptoms of Prostate Cancer | pre-intervention (T1), post-intervention (8 weeks after T1)
  The investigators will assess symptoms associated with prostate cancer and its treatment with the German version of the 'Expanded Prostate Cancer Index Composite' (EPIC-26, [Wei et al., 2000]). The EPIC-26 is a self-reported measure to assess patient function and distress after prostate cancer treatment. It covers multiple health-related quality of life (HRQOL) domains, namely urinary (incontinence and irritative/obstructive), bowel, sexual, and hormonal functionality. Each of these domains are assessed in terms of their function and bother and summarized into domain summary scores. The higher the EPIC-26 score (maximum 100 points), the better the patient's assessment of functionality in the dimension covered. This scale will only be completed by prostate cancer patients.
Treatment Expectancy and Rational Credibility | pre-intervention (T1)
  In order to assess prostate cancer patients' expectancy and the perceived credibility of the WINGS-IP1 Smartphone Application the investigators will use the 'Credibility Expectancy Questionnaire' (CEQ, [Devilly & Borkovec, 2000]). A total of six items are rated on a 1-9 or a 0%-100% scale, depending upon the item. Higher scores refer to higher expectancy and higher credibility. This scale will only be completed by prostate cancer patients.
Hospital Record Data on Prostate Cancer Symptoms | six months post-prostatectomy
  In addition, the 'Expanded Prostate Cancer Index Composite' (EPIC-26, [Wei et al., 2000]) will be assessed in prostate cancer patients six months post-prostatectomy as part of the clinical standard procedures at the University Hospital Basel. Hence, instead of a follow-up assessment 12 weeks after T1, the investigators will retrieve prostate cancer patients' EPIC-26 data from hospital records entered during the standard six months post-prostatectomy follow-up.

OTHER OUTCOMES:
Internet Self-Efficacy Scale | pre-intervention
  In order to measure patients' beliefs in their capabilities to use the German version of the Internet and Internet-based programs the investigators will use the 'Internet Self-efficacy Scale' (ISS, [Eastin & LaRose, 2006]). The ISS is a self-report measure, including 10 items rated on a seven-point Likert-scale ranging from 1 = "strongly disagree" to 7 = "strongly agree". For the purpose of this study, the investigators will translate the ISS into German. This scale will be completed by prostate cancer patients and their supporters.
Reported Use Frequency Post-Intervention | post-intervention (after 8 weeks)
  The investigators will ask patients and their supporters to declare how often they have used the WINGS Smartphone Application during the eight-week intervention phase (e.g., daily, every other day, three times a week, twice a week, once a week, less than once a week).
Reported Use Frequency Follow-up | follow-up (after 12 weeks)
  The investigators will ask patients and their supporters to declare how often they have used the WINGS Smartphone Application during the eight-week intervention phase (e.g., daily, every other day, three times a week, twice a week, once a week, less than once a week).
Reported Number of Supporters Contacted by Patients Post-Intervention | post-intervention (after 8 weeks)
  The investigators will ask patients to declare how many supporters they have contacted via WINGS Smartphone Application.
Reported Number of Supporters Contacted by Patients Follow-up | follow-up (after 12 weeks)
  The investigators will ask patients to declare how many supporters they have contacted via WINGS Smartphone Application.
Number of Supporters per Patient Post-Intervention in WINGS Smartphone Application | post-intervention (after 8 weeks)
  The investigators will extract the number of supporters per individual patient directly from the WINGS Smartphone Application.
Number of Supporters per Patient Follow-up WINGS Smartphone Application | follow-up (after 12 weeks)
  The investigators will extract the number of supporters per individual patient directly from the WINGS Smartphone Application.
Reported Psycho-Oncological Consultation Uptake Post-Intervention | post-intervention (after 8 weeks)
  The investigators will ask prostate cancer patients if they had taken up psycho-oncological consultation before or after their prostatectomy.
Psycho-Oncological Consultation Uptake Post-Intervention in Hospital Records | post-intervention (after 8 weeks)
  The investigators will consult hospital records to check whether patients have had any psycho-oncological consultations.
Reported Psycho-Oncological Consultation Uptake Follow-up | follow-up (after 12 weeks)
  The investigators will ask prostate cancer patients if they had taken up psycho-oncological consultation before or after their prostatectomy.
Psycho-Oncological Consultation Uptake Follow-up in Hospital Records | follow-up (after 12 weeks)
  The investigators will consult hospital records to check whether patients have had any psycho-oncological consultations.
Report of Adverse Event (AE) and/or Device Deficiency (DD) | through study completion, an average of 3 months
  The investigators will ask prostate cancer patients and their supporters to report any Adverse Events (AEs) in free text format.
Report of Device Deficiency (DD) | through study completion, an average of 3 months
  The investigators will ask prostate cancer patients and their supporters to report any Device Deficiencies (DDs) in free text format.
General Feedback Post-Intervention | post-intervention (after 8 weeks)
  The investigators will ask prostate cancer patients and their supporters to provide general feedback on the WINGS Smartphone Application.
General Feedback Follow-up | follow-up (after 12 weeks)
  The investigators will ask prostate cancer patients and their supporters to provide general feedback on the WINGS Smartphone Application.
Adverse Event (AE) and/or Device Deficiency (DD) Assessed by Investigators | through study completion, an average of 3 months
  The investigators will adequately assess any undesired side effects of the intervention and document the rate of adverse events in general, considering reports of adverse events or device deficiency by prostate cancer patients and supporters. The investigators will also monitor (severe) Adverse Events (AEs) relating to participants' disease progression, including (but not limited to) death and hospitalization. AEs will be designated and managed according to ICH-GCP E6 (International Conference on Harmonization (ICH), 2016). All AEs that occur during the study will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Meinlschmidt, Prof. Dr., Principal Investigator — University Hospital Basel, Basel Switzerland; Rainer Schaefert, Prof. Dr., Principal Investigator — University Hospital Basel, Basel Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller SM, Hudson SV, Hui SK, Diefenbach MA, Fleisher L, Raivitch S, Belton T, Roy G, Njoku A, Scarpato J, Viterbo R, Buyyounouski M, Denlinger C, Miyamoto C, Reese A, Baman J. Development and preliminary testing of PROGRESS: a Web-based education program for prostate cancer survivors transitioning from active treatment. J Cancer Surviv. 2015 Sep;9(3):541-53. doi: 10.1007/s11764-015-0431-5. Epub 2015 Feb 20. PMID 25697335
- [Background] Bacon CG, Giovannucci E, Testa M, Glass TA, Kawachi I. The association of treatment-related symptoms with quality-of-life outcomes for localized prostate carcinoma patients. Cancer. 2002 Feb 1;94(3):862-71. doi: 10.1002/cncr.10248. PMID 11857323
- [Background] Badger TA, Segrin C, Figueredo AJ, Harrington J, Sheppard K, Passalacqua S, Pasvogel A, Bishop M. Who benefits from a psychosocial counselling versus educational intervention to improve psychological quality of life in prostate cancer survivors? Psychol Health. 2013;28(3):336-54. doi: 10.1080/08870446.2012.731058. Epub 2012 Oct 9. PMID 23045995
- [Background] Bennett G, Badger TA. Depression in men with prostate cancer. Oncol Nurs Forum. 2005 May 10;32(3):545-56. doi: 10.1188/05.ONF.545-556. PMID 15897931
- [Background] Chipperfield K, Fletcher J, Millar J, Brooker J, Smith R, Frydenberg M, Oh T, Burney S. Factors associated with adherence to physical activity guidelines in patients with prostate cancer. Psychooncology. 2013 Nov;22(11):2478-86. doi: 10.1002/pon.3310. Epub 2013 Jun 7. PMID 23749430
- [Background] Lintz K, Moynihan C, Steginga S, Norman A, Eeles R, Huddart R, Dearnaley D, Watson M. Prostate cancer patients' support and psychological care needs: Survey from a non-surgical oncology clinic. Psychooncology. 2003 Dec;12(8):769-83. doi: 10.1002/pon.702. PMID 14681951
- [Background] Wootten AC, Burney S, Foroudi F, Frydenberg M, Coleman G, Ng KT. Psychological adjustment of survivors of localised prostate cancer: investigating the role of dyadic adjustment, cognitive appraisal and coping style. Psychooncology. 2007 Nov;16(11):994-1002. doi: 10.1002/pon.1159. PMID 17278153
- [Background] Siegel SD, Molton I, Penedo FJ, Llabre MM, Kinsinger DP, Traeger L, Schneiderman N, Antoni MH. Interpersonal sensitivity, partner support, patient-physician communication, and sexual functioning in men recovering from prostate carcinoma. J Pers Assess. 2007 Dec;89(3):303-9. doi: 10.1080/00223890701629847. PMID 18001230
- [Background] Wittmann D, Carolan M, Given B, Skolarus TA, An L, Palapattu G, Montie JE. Exploring the role of the partner in couples' sexual recovery after surgery for prostate cancer. Support Care Cancer. 2014 Sep;22(9):2509-15. doi: 10.1007/s00520-014-2244-x. Epub 2014 Apr 13. PMID 24728619
- [Background] Karakiewicz PI, Bhojani N, Neugut A, Shariat SF, Jeldres C, Graefen M, Perrotte P, Peloquin F, Kattan MW. The effect of comorbidity and socioeconomic status on sexual and urinary function and on general health-related quality of life in men treated with radical prostatectomy for localized prostate cancer. J Sex Med. 2008 Apr;5(4):919-927. doi: 10.1111/j.1743-6109.2007.00741.x. PMID 18371045
- [Background] Couper JW, Bloch S, Love A, Duchesne G, Macvean M, Kissane DW. The psychosocial impact of prostate cancer on patients and their partners. Med J Aust. 2006 Oct 16;185(8):428-32. doi: 10.5694/j.1326-5377.2006.tb00640.x. PMID 17137432
- [Background] Wood A, Barden S, Terk M, Cesaretti J. Prostate cancer: the influence of stigma on quality of life and relationship satisfaction for survivors and their partners. J Psychosoc Oncol. 2019 May-Jun;37(3):350-366. doi: 10.1080/07347332.2018.1489442. Epub 2018 Dec 22. PMID 30580663
- [Background] Lambert SD, Girgis A, Lecathelinais C, Stacey F. Walking a mile in their shoes: anxiety and depression among partners and caregivers of cancer survivors at 6 and 12 months post-diagnosis. Support Care Cancer. 2013 Jan;21(1):75-85. doi: 10.1007/s00520-012-1495-7. Epub 2012 Jun 3. PMID 22661096
- [Background] Merz EL, Malcarne VL, Ko CM, Sadler M, Kwack L, Varni JW, Sadler GR. Dyadic concordance among prostate cancer patients and their partners and health-related quality of life: does it matter? Psychol Health. 2011 Jun;26(6):651-66. doi: 10.1080/08870441003721251. Epub 2011 Jul 11. PMID 20680885
- [Background] Segrin C, Badger TA, Harrington J. Interdependent psychological quality of life in dyads adjusting to prostate cancer. Health Psychol. 2012 Jan;31(1):70-9. doi: 10.1037/a0025394. Epub 2011 Sep 5. PMID 21895374
- [Background] Kim Y, Carver CS, Ting A, Cannady RS. Passages of cancer caregivers' unmet needs across 8 years. Cancer. 2020 Oct 15;126(20):4593-4601. doi: 10.1002/cncr.33053. Epub 2020 Aug 8. PMID 32770755
- [Background] Song L, Rini C, Ellis KR, Northouse LL. Appraisals, perceived dyadic communication, and quality of life over time among couples coping with prostate cancer. Support Care Cancer. 2016 Sep;24(9):3757-65. doi: 10.1007/s00520-016-3188-0. Epub 2016 Apr 2. PMID 27039207
- [Background] Berkman LF, Glass T, Brissette I, Seeman TE. From social integration to health: Durkheim in the new millennium. Soc Sci Med. 2000 Sep;51(6):843-57. doi: 10.1016/s0277-9536(00)00065-4. PMID 10972429
- [Background] Carpenter KM, Fowler JM, Maxwell GL, Andersen BL. Direct and buffering effects of social support among gynecologic cancer survivors. Ann Behav Med. 2010 Feb;39(1):79-90. doi: 10.1007/s12160-010-9160-1. PMID 20151235
- [Background] Rivera Rivera JN, Burris JL. A Systematic Literature Review and Head-to-Head Comparison of Social Support and Social Constraint in Relation to the Psychological Functioning of Cancer Survivors. Ann Behav Med. 2020 Feb 21;54(3):176-192. doi: 10.1093/abm/kaz037. PMID 31581293
- [Background] Sauer C, Weis J, Faller H, Junne F, Honig K, Bergelt C, Hornemann B, Stein B, Teufel M, Goerling U, Erim Y, Geiser F, Niecke A, Senf B, Weber D, Maatouk I. Impact of social support on psychosocial symptoms and quality of life in cancer patients: results of a multilevel model approach from a longitudinal multicenter study. Acta Oncol. 2019 Sep;58(9):1298-1306. doi: 10.1080/0284186X.2019.1631471. Epub 2019 Jul 9. PMID 31284793
- [Background] Mehnert A, Lehmann C, Graefen M, Huland H, Koch U. Depression, anxiety, post-traumatic stress disorder and health-related quality of life and its association with social support in ambulatory prostate cancer patients. Eur J Cancer Care (Engl). 2010 Nov;19(6):736-45. doi: 10.1111/j.1365-2354.2009.01117.x. PMID 19832893
- [Background] McCaughan E, Curran C, Northouse L, Parahoo K. Evaluating a psychosocial intervention for men with prostate cancer and their partners: Outcomes and lessons learned from a randomized controlled trial. Appl Nurs Res. 2018 Apr;40:143-151. doi: 10.1016/j.apnr.2018.01.008. Epub 2018 Jan 31. PMID 29579490
- [Background] Docherty A, Brothwell CP, Symons M. The impact of inadequate knowledge on patient and spouse experience of prostate cancer. Cancer Nurs. 2007 Jan-Feb;30(1):58-63. doi: 10.1097/00002820-200701000-00011. PMID 17235222
- [Background] Bailey DE Jr, Wallace M, Mishel MH. Watching, waiting and uncertainty in prostate cancer. J Clin Nurs. 2007 Apr;16(4):734-41. doi: 10.1111/j.1365-2702.2005.01545.x. PMID 17402955
- [Background] Banerjee S, Califano R, Corral J, de Azambuja E, De Mattos-Arruda L, Guarneri V, Hutka M, Jordan K, Martinelli E, Mountzios G, Ozturk MA, Petrova M, Postel-Vinay S, Preusser M, Qvortrup C, Volkov MNM, Tabernero J, Olmos D, Strijbos MH. Professional burnout in European young oncologists: results of the European Society for Medical Oncology (ESMO) Young Oncologists Committee Burnout Survey. Ann Oncol. 2017 Jul 1;28(7):1590-1596. doi: 10.1093/annonc/mdx196. PMID 28449049
- [Background] Penedo FJ, Fox RS, Oswald LB, Moreno PI, Boland CL, Estabrook R, McGinty HL, Mohr DC, Begale MJ, Dahn JR, Flury SC, Perry KT, Kundu SD, Yanez B. Technology-Based Psychosocial Intervention to Improve Quality of Life and Reduce Symptom Burden in Men with Advanced Prostate Cancer: Results from a Randomized Controlled Trial. Int J Behav Med. 2020 Oct;27(5):490-505. doi: 10.1007/s12529-019-09839-7. PMID 31898309
- [Background] Bouchard LC, Yanez B, Dahn JR, Flury SC, Perry KT, Mohr DC, Penedo FJ. Brief report of a tablet-delivered psychosocial intervention for men with advanced prostate cancer: Acceptability and efficacy by race. Transl Behav Med. 2019 Jul 16;9(4):629-637. doi: 10.1093/tbm/iby089. PMID 30285186
- [Background] Handley NR, Wen KY, Gomaa S, Brassil K, Shimada A, Leiby B, Jackson L, McMorris M, Calvaresi A, Dicker AP. A Pilot Feasibility Study of Digital Health Coaching for Men With Prostate Cancer. JCO Oncol Pract. 2022 Jul;18(7):e1132-e1140. doi: 10.1200/OP.21.00712. Epub 2022 Apr 8. PMID 35394806
- [Background] Agochukwu NQ, Skolarus TA, Wittmann D. Telemedicine and prostate cancer survivorship: a narrative review. Mhealth. 2018 Oct 8;4:45. doi: 10.21037/mhealth.2018.09.08. eCollection 2018. PMID 30505843
- [Background] Pai HH, Lau F. Web-based electronic health information systems for prostate cancer patients. Can J Urol. 2005 Jun;12(3):2700-9. PMID 16011818
- [Background] Campbell LC, Keefe FJ, McKee DC, Waters SJ, Moul JW. Masculinity beliefs predict psychosocial functioning in African American prostate cancer survivors. Am J Mens Health. 2012 Sep;6(5):400-8. doi: 10.1177/1557988312450185. Epub 2012 Jun 11. PMID 22691305
- [Background] Wood AW, Barden S, Terk M, Cesaretti J. The influence of stigma on the quality of life for prostate cancer survivors. J Psychosoc Oncol. 2017 Jul-Aug;35(4):451-467. doi: 10.1080/07347332.2017.1307896. Epub 2017 Mar 20. PMID 28318410
- [Background] Lyon AR, Pullmann MD, Jacobson J, Osterhage K, Achkar MA, Renn BN, Munson SA, Arean PA. Assessing the Usability of Complex Psychosocial Interventions: The Intervention Usability Scale. Implement Res Pract. 2021 Jan-Dec;2:2633489520987828. doi: 10.1177/2633489520987828. Epub 2021 Feb 8. PMID 35601889
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Pressler SJ, Subramanian U, Perkins SM, Gradus-Pizlo I, Kareken D, Kim J, Ding Y, Sauve MJ, Sloan R. Measuring depressive symptoms in heart failure: validity and reliability of the patient health questionnaire-8. Am J Crit Care. 2011 Mar;20(2):146-52. doi: 10.4037/ajcc2010931. Epub 2010 Apr 8. PMID 20378777
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Staples LG, Dear BF, Gandy M, Fogliati V, Fogliati R, Karin E, Nielssen O, Titov N. Psychometric properties and clinical utility of brief measures of depression, anxiety, and general distress: The PHQ-2, GAD-2, and K-6. Gen Hosp Psychiatry. 2019 Jan-Feb;56:13-18. doi: 10.1016/j.genhosppsych.2018.11.003. Epub 2018 Nov 22. PMID 30508772
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Fife BL, Wright ER. The dimensionality of stigma: a comparison of its impact on the self of persons with HIV/AIDS and cancer. J Health Soc Behav. 2000 Mar;41(1):50-67. PMID 10750322
- [Background] Eichhorn S, Mehnert A, Stephan M. [German Version of the Social Impact Scale (SIS-D)--Pilot Testing of an Instrument for Measuring Experienced Stigmatization in a Sample of Cancer Patients]. Psychother Psychosom Med Psychol. 2015 May;65(5):183-90. doi: 10.1055/s-0034-1398523. Epub 2015 Mar 20. German. PMID 25794353
- [Background] Dalgard OS, Dowrick C, Lehtinen V, Vazquez-Barquero JL, Casey P, Wilkinson G, Ayuso-Mateos JL, Page H, Dunn G; ODIN Group. Negative life events, social support and gender difference in depression: a multinational community survey with data from the ODIN study. Soc Psychiatry Psychiatr Epidemiol. 2006 Jun;41(6):444-51. doi: 10.1007/s00127-006-0051-5. Epub 2006 Mar 29. PMID 16572275
- [Background] Toussaint A, Murray AM, Voigt K, Herzog A, Gierk B, Kroenke K, Rief W, Henningsen P, Lowe B. Development and Validation of the Somatic Symptom Disorder-B Criteria Scale (SSD-12). Psychosom Med. 2016 Jan;78(1):5-12. doi: 10.1097/PSY.0000000000000240. PMID 26461855
- [Background] Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology. 2000 Dec 20;56(6):899-905. doi: 10.1016/s0090-4295(00)00858-x. PMID 11113727
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Berry N, Bucci S, Lobban F. Use of the Internet and Mobile Phones for Self-Management of Severe Mental Health Problems: Qualitative Study of Staff Views. JMIR Ment Health. 2017 Nov 1;4(4):e52. doi: 10.2196/mental.8311. PMID 29092809